CLINICAL TRIAL: NCT05521347
Title: Graduate Program in Department of Exercise Health Science, National Taiwan University of Sport
Brief Title: Caffeine Supplementation Improves the Cognitive Abilities and Shooting Performance of Trained E-sports Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Associate Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 111-1
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Caffeine; Placebo
Keywords: caffeine; reaction time
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine (Experimental): capsules with 3 mg/kg of caffeine
  Interventions: Behavioral: caffeine
- placebo (Placebo Comparator): The placebo capsule contained flour
  Interventions: Behavioral: caffeine

INTERVENTIONS:
Behavioral: caffeine — we employed a randomized crossover design to divide participants into a caffeine trial (CAF) and a placebo trial (PL). The CAF group took capsules with 3 mg/kg of caffeine, whereas the PL group took a placebo capsule. After a 1-h rest, the Stroop task, visual search ability test, and the shooting ability test were conducted.

SUMMARY:
Purpose: investigators explored the effect of 3 mg/kg of caffeine supplementation on the cognitive ability and shooting performance of trained e-sports players. Methods: investigators recruited nine e-sports players who had received professional training in e-sports and had won at least eighth place in national-level e-sports shooting competitions. After performing three to five familiarization tests, investigators employed a randomized crossover design to divide participants into a caffeine trial (CAF) and a placebo trial (PL). The CAF group took capsules with 3 mg/kg of caffeine, whereas the PL group took a placebo capsule. After a 1-h rest, the Stroop task, visual search ability test, and the shooting ability test were conducted.

ELIGIBILITY:
Inclusion Criteria:

* had experience with national competitions and regularly underwent training in first-person shooters

Exclusion Criteria:

* no experience with national competitions and regularly underwent training in first-person shooters
* have any diseases affecting the heart, bones, and joints or diseases that preclude exercise

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male subjects
Enrollment: 9 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Stroop task | 1 hour after intervention
  The color-word Stroop task and visual search test were conducted using Psych/Lab for Windows. The reaction time (millisecond) were recorded.
visual search test | 1 hour after intervention
  A total of 80 search displays were presented in 5 minutes. In each display, 5, 10, 15, or 20 -Tests were presented. The reaction time (millisecond) were recorded.

SECONDARY OUTCOMES:
aim trainer | 1 hour after intervention
  Participants used the mouse to shoot the electronic targets on the computer screen. The completed time (second) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

DOCUMENTS (1):
  • Study Protocol (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT05521347/Prot_000.pdf